CLINICAL TRIAL: NCT06698198
Title: Safety and Immunogenicity of a Pneumococcal Conjugate Vaccine Candidate in Healthy Adults (19-49 Years)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PSK00007; PSK00007 (Other: Sanofi); U1111-1210-0812 (Registry Identifier: ICTRP)
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-08

CONDITIONS: Pneumococcal Immunization
MeSH Terms: interventions — Pneumococcal Vaccines; 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Group 1: Pneumococcal Conjugate Vaccine (PCV) SP0202-I (Experimental): Participants will receive 1 intramuscular injection of PCV formulation SP0202-I
  Interventions: Biological: Pneumococcal Conjugate Vaccine
- Group 2: Pneumococcal Conjugate Vaccine (PCV) SP0202-II (Experimental): Participants will receive 1 intramuscular injection of PCV formulation SP0202-II
  Interventions: Biological: Pneumococcal Conjugate Vaccine
- Group 3: Pneumococcal Conjugate Vaccine (PCV) SP0202-III (Experimental): Participants will receive 1 intramuscular injection of PCV formulation SP0202-III
  Interventions: Biological: Pneumococcal Conjugate Vaccine
- Group 4: Pneumococcal Conjugate Vaccine (PCV) SP0202-IV (Experimental): Participants will receive 1 intramuscular injection of PCV formulation SP0202-IV
  Interventions: Biological: Pneumococcal Conjugate Vaccine
- Group 5: Prevnar 13® (Active Comparator)
  Interventions: Biological: Prevnar 13®

INTERVENTIONS:
Biological: Pneumococcal Conjugate Vaccine — Suspension for Intramuscular injection
  Arms: Group 1: Pneumococcal Conjugate Vaccine (PCV) SP0202-I; Group 2: Pneumococcal Conjugate Vaccine (PCV) SP0202-II; Group 3: Pneumococcal Conjugate Vaccine (PCV) SP0202-III; Group 4: Pneumococcal Conjugate Vaccine (PCV) SP0202-IV
Biological: Prevnar 13® — Suspension for Intramuscular injection
  Arms: Group 5: Prevnar 13®

SUMMARY:
This was a Phase I, randomized, active-controlled, observer-blinded, multi-center study to assess the safety and the immunogenicity of 4 Pneumococcal Conjugate Vaccines (PCV) candidates in parallel with Prevnar 13, in Healthy Adults (19-49 years) in the United States.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 19 to 49 years on the day of inclusion ("19 to 49 years" means from the day of the 19th birthday to the day before the 50th birthday)
* Informed Consent Form (ICF) has been signed and dated
* Able to attend all scheduled visits and to comply with all trial procedures
* Body mass index within the range of 18.5 and 29.9 kg/m2

Exclusion Criteria:

* Subject is pregnant, or lactating, or of childbearing potential and not using an effective method of contraception or abstinence from at least 4 weeks prior to vaccine injection until at least 4 weeks after injection. To be considered of non-childbearing potential, a female must be pre-menarche, or post-menopausal for at least 1 year, or surgically sterile.
* Participation at the time of study enrollment (or in the 4 weeks preceding the trial vaccination) or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 4 weeks preceding the trial vaccination or planned receipt of any vaccine in the 4 weeks following trial injection, except for influenza vaccination, which may be received at least 2 weeks before SP0202 or Prevnar 13 injection.
* Previous vaccination against S. pneumoniae with either a pneumococcal conjugate vaccine (PCV) or a Pneumococcal polysaccharide vaccines (PPSV).
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 19 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 175 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Occurrence of unsolicited systemic AEs reported in the 30 minutes after injection | Up to 30 minutes post-vaccination
  Occurrence of any unsolicited (spontaneously reported) systemic Adverse Events (AEs) reported in the 30 minutes after injection of a SP0202 formulation or Prevnar 13.
Occurrence of solicited injection site and systemic reactions | Up to 7 days post-vaccination
  Number of participants reporting solicited injection site reactions (pain, redness, swelling) and solicited systemic reactions (pyrexia, headache, malaise, myalgia, arthralgia, chills)
Occurrence of unsolicited (spontaneously reported) AEs up to 30 days after injection | Up to 30 days after vaccination
  Occurrence of unsolicited (spontaneously reported) Adverse Events (AEs) up to 30 days after injection of a SP0202 formulation or Prevnar 13.
Serotype-specific immunoglobulin type G (IgG) concentrations | Up to 30 days after vaccination
  Geometric Mean (GM) of serotype-specific IgG concentrations for all pneumococcal serotypes included in the Pneumococcal Conjugate Vaccine (PCV) formulations, as measured by electro-chemiluminescence (ECL) assay
Serotype-specific opsonophagocytic activity (OPA) titers | Up to 30 days after vaccination
  GM of serotype-specific OPA titers for all pneumococcal serotypes included in the Pneumococcal Conjugate Vaccine (PCV) formulations, as determined by multiplex opsonophagocytic assay (MOPA)

SECONDARY OUTCOMES:
Serotype-specific IgG concentrations ratio (post/pre-vaccination) | Up to 30 days after vaccination
  GM of serotype-specific IgG concentrations ratio (post-/pre-vaccination) for each pneumococcal serotypes included in the Pneumococcal Conjugate Vaccine (PCV) formulations, as measured by ECL assay
≥ 4-fold serotype-specific IgG concentrations increase | Up to 30 days after vaccination
  Percentage of participants with ≥ 4-fold serotype-specific IgG concentrations increase from baseline to 1 month post-vaccination for each pneumococcal serotypes included in the Pneumococcal Conjugate Vaccine (PCV) formulations, as measured by ECL
Serotype-specific OPA titers ratio (post/pre-vaccination) | Up to 30 days after vaccination
  GM of serotype-specific OPA titers ratio (post-/pre-vaccination) for each pneumococcal serotypes included in the Pneumococcal Conjugate Vaccine (PCV) formulations, as determined by MOPA
≥ 4-fold serotype-specific OPA titers increase | Up to 30 days after vaccination
  Percentage of participants with ≥ 4-fold serotype-specific IgG concentrations increase from baseline to post-vaccination for each pneumococcal serotypes included in the Pneumococcal Conjugate Vaccine (PCV) formulations, as determined by MOPA

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (2):
- United States (2):
  - Investigational Site Number: 0002, Metairie, Louisiana
  - Investigational Site Number: 0001, Newark, New Jersey

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org